CLINICAL TRIAL: NCT07155018
Title: Effectiveness of Micro-Osteoperforations (MOPs) in Accelerating Maxillary Canine Retraction in Angle Class I Malocclusion: A Randomized Controlled Trial.
Brief Title: Micro-Osteoperforations to Accelerate Maxillary Canine Retraction in Class I Malocclusion
Acronym: MOPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DuongThaoTrangCtump; IRB-164- (Registry Identifier: Ethics Committee of Can Tho University of Medicine and Pharmacy)
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Malocclusion, Angle Class I
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: This is a single-blinded, split-mouth randomized controlled trial. Each participant received both interventions: on one side of the maxillary arch, micro-osteoperforations (MOPs) were performed distal to the canine, while the contralateral side served as the control with conventional retraction. Outcomes were measured within the same patient, reducing inter-individual variability.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor was blinded to the intervention allocation. Patients and treating clinicians were aware of the intervention side, but the examiner performing digital measurements and statistical analysis did not know which side received MOPs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Micro-osteoperforations (Experimental): On the experimental side, micro-osteoperforations (MOPs) were performed distal to the maxillary canine under local anesthesia using the Excellerator RT device. Three perforations, each 1.5 mm in diameter and 5 mm deep, were created in the attached gingiva. Canine retraction was then carried out using miniscrew anchorage and NiTi closed-coil springs.
  Interventions: Procedure: Micro-osteoperforations (MOPs)
- Control: Conventional Retraction (Active Comparator): On the control side, maxillary canine retraction was performed using miniscrew anchorage and NiTi closed-coil springs without any micro-osteoperforations. The mechanics were identical to the experimental side to ensure comparability.
  Interventions: Procedure: Conventional Canine Retraction

INTERVENTIONS:
Procedure: Micro-osteoperforations (MOPs) — Maxillary canine retraction with miniscrew anchorage and NiTi closed-coil springs, without micro-osteoperforations.
  Arms: Experimental: Micro-osteoperforations
Procedure: Conventional Canine Retraction — Maxillary canine retraction with miniscrew anchorage and NiTi closed-coil springs, without micro-osteoperforations
  Arms: Control: Conventional Retraction

SUMMARY:
This single-blinded, split-mouth randomized controlled trial investigates whether micro-osteoperforations (MOPs) can accelerate maxillary canine retraction in orthodontic patients requiring bilateral premolar extraction. The study also evaluates postoperative pain levels using the Visual Analog Scale at 1, 3, and 7 days.

DETAILED DESCRIPTION:
MOPs are a flapless, minimally invasive surgical technique that stimulates bone remodeling and may reduce orthodontic treatment time. In this trial, one side of each patient receives MOPs while the contralateral side serves as control. Canine retraction is performed using miniscrews, power arms, and NiTi coil springs. Outcomes include the rate of canine movement over 16 weeks and pain assessment using VAS.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-25 years
* Patients requiring bilateral extraction of maxillary first premolars as part of orthodontic treatment
* Angle Class I molar relationship
* No previous orthodontic treatment

Exclusion Criteria:

* History of craniofacial trauma or congenital anomalies
* Systemic or bone-related diseases
* Current smoking
* Use of medications affecting bone metabolism

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of Maxillary Canine Retraction | Baseline, 4, 8, 12, and 16 weeks
  Distance of maxillary canine retraction measured on 3D digital dental models using intraoral scanning.

SECONDARY OUTCOMES:
Pain Level (VAS Score) | Day 1, Day 3, Day 7 after intervention
  atient-reported pain intensity measured using a 10-cm Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Lam Nguyen Le, Ph.D.DDS, Study Chair — Department of Pediatrics Dentistry and Orthodontics, Faculty of Odonto- Stomatology, Can Tho University of Medicine and Pharmacy, Can Tho City, Vietnam
Locations (1):
- Can Tho University Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study has a small sample size and the data may compromise patient confidentiality.